CLINICAL TRIAL: NCT06746610
Title: Screening and Molecular Diagnosis-based Individualized Precision Management of Monogenic Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Hua Shu, Attending Physician, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB2022-YX-164-01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Monogenic Diabetes
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Monogenic Diabetes Genetic Screening and Molecular Diagnosis (Other)
  Interventions: Diagnostic Test: Genetic Screening for Monogenic Diabetes

INTERVENTIONS:
Diagnostic Test: Genetic Screening for Monogenic Diabetes — This intervention involves genetic testing for monogenic diabetes (MDM) in recruited participants. The testing includes either a panel test specifically targeting genes associated with monogenic diabetes or whole exome sequencing (WES) to comprehensively identify genetic variants linked to MDM.
  Precise diagnosis and treatmen：
  1. The clinical trial of individualized treatment was carried out for the individuals with diabetes with HNF1A mutation.
  2. The research team will closely follow up individuals with GCK mutation diabetes after suspending the current hypoglycemic drugs, and evaluate their clinical glucose metabolism related indicators.
  3. Observe the dosage of sulfonylurea drugs used in individuals with different disease course and pancreatic function, and observe the impact of disease course and pancreatic function on the success rate of oral drug replacement.

SUMMARY:
The goal of this observational study is to establish a registry, screening, and individualized management platform for patients with monogenic diabetes mellitus(MDM) using internet-based and mobile application software. The main questions it aims to answer are:

* What are the genetic mutations causing MDM in China (genetic landscape)?
* How effective and safe is the individualized, molecular-diagnosis-based management platform for MDM in improving patient outcomes?

Participants will:

* Register in the MDM platform via mobile app or internet-based software
* Undergo genetic screening for MDM diagnosis
* Participate in follow-up visits for individualized management and monitoring of blood glucose control and outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes patients who developed before 25 years old; Or they were diagnosed with diabetes before the age of 35, and two or more immediate relatives were diagnosed with diabetes before the age of 45;
2. Body mass index (BMI) at diagnosis < 28 kg/m2;
3. Anti glutamic acid decarboxylase antibody (GAD Ab), anti islet cell antibody (ICA Ab), and anti insulin autoantibody (IAA Ab) were all negative;

Exclusion Criteria:

1. Secondary diabetes patients with other endocrine diseases, such as hyperthyroidism or hypothyroidism, hyperparathyroidism or hypothyroidism, acromegaly, Cushing's syndrome, autoimmune multiple endocrine diseases, etc.;
2. Systemic use of corticosteroids, immunosuppressants, and other drugs within the past 6 months;
3. Patients with malignant tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Genetic landscape of monogenic diabetes mellitus in China | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China